CLINICAL TRIAL: NCT06990295
Title: Effects of Focused Ultrasound Spleen Neuromodulation on Inflammatory Cytokine Levels in Patients With Septic Shock: A Randomized Controlled Pilot Trial
Brief Title: Focused Ultrasound Spleen Stimulation and Inflammation in Septic Shock
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Wannan Medical College (Other)
Collaborators: Wuhu City Second People's Hospital (Other)
Responsible Party: Principal Investigator, Qiancheng Xu, Principal Investigator, First Affiliated Hospital of Wannan Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202580
Record Dates: First submitted 2025-05-18; First posted 2025-05-25 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Septic Shock; Inflammatory Cytokines; Spleen Neuromodulation; Focused Ultrasound; Critical Care
Keywords: Septic Shock; Focused Ultrasound; Spleen Neuromodulation; Inflammatory Cytokines; Critical Care; Immune Modulation; Pilot Study
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Focused Ultrasound Spleen Neuromodulation Group (Experimental): Patients receive standard septic shock care plus twice-daily non-invasive focused ultrasound stimulation over the spleen for five consecutive days, using a portable ultrasound neuromodulation device.
  Interventions: Procedure: Focused Ultrasound Spleen Neuromodulation
- Control Group (No Intervention): Patients receive standard care for septic shock according to current clinical guidelines, without focused ultrasound spleen stimulation.

INTERVENTIONS:
Procedure: Focused Ultrasound Spleen Neuromodulation — A portable focused ultrasound device is used to stimulate the spleen area under real-time imaging guidance. Each session lasts approximately 20 minutes, repeated twice daily for five days.
  Arms: Focused Ultrasound Spleen Neuromodulation Group

SUMMARY:
This study evaluates the safety and effectiveness of focused ultrasound spleen neuromodulation in patients with septic shock, a life-threatening condition characterized by excessive inflammation and organ dysfunction. The primary objective is to determine whether non-invasive, focused ultrasound stimulation of the spleen can reduce circulating inflammatory cytokine levels in this patient population.

Eligibility Criteria:

Adults aged 18 years or older Diagnosed with septic shock and admitted to the ICU within 24 hours Expected to require intensive care for at least 72 hours

Study Protocol:

Participants will be randomly assigned to one of two groups:

Intervention Group: Will receive standard septic shock care plus twice-daily focused ultrasound stimulation over the spleen for five days, using a portable device.

Control Group: Will receive standard septic shock care alone. Blood samples will be collected at baseline, Day 3, and Day 5 to measure inflammatory cytokine levels, including TNF-α, IL-1β, IL-6, and IL-10. Additional assessments will include lymphocyte subpopulations, organ function scores, ICU length of stay, 28-day mortality, and adverse events.

Outcome Measures:

Primary: Change in levels of inflammatory cytokines on Day 3 and Day 5. Secondary: Changes in organ function (SOFA score), ICU length of stay, 28-day survival, and safety/tolerability of the intervention.

DETAILED DESCRIPTION:
This randomized, controlled pilot study investigates the safety and efficacy of focused ultrasound neuromodulation of the spleen in adult patients diagnosed with septic shock. Participants will be randomized into two groups: one receiving standard of care and the other receiving additional targeted spleen stimulation via focused ultrasound. The intervention involves twice-daily sessions over five days, utilizing a portable device designed to deliver precise, non-invasive ultrasound energy to the splenic region. The rationale for targeting the spleen stems from its role in immunomodulation, particularly in the regulation of inflammatory cytokines involved in septic shock pathophysiology.

Blood samples will be systematically collected at baseline, Day 3, and Day 5 to quantify serum levels of key inflammatory cytokines, including tumor necrosis factor-alpha (TNF-α), interleukin-1 beta (IL-1β), interleukin-6 (IL-6), and interleukin-10 (IL-10), using validated immunoassays. In addition, lymphocyte subpopulations will be analyzed via flow cytometry to assess immune cell dynamics. Organ dysfunction will be evaluated using the Sequential Organ Failure Assessment (SOFA) score at specified time points to monitor changes in organ status. Data on ICU length of stay and 28-day mortality will be collected to evaluate clinical outcomes. Adverse events related to the intervention will be documented to assess safety and tolerability.

By investigating the immunomodulatory effects of focused ultrasound spleen neuromodulation, this study aims to establish preliminary safety and efficacy data for a potentially transformative therapeutic modality in septic shock management.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, regardless of sex
* Diagnosed with septic shock according to Sepsis-3 criteria: Sequential Organ Failure Assessment (SOFA) score ≥ 2 and requiring vasopressor support to maintain a mean arterial pressure (MAP) ≥ 65 mmHg.
* Admitted to the ICU within 24 hours of septic shock diagnosis
* Expected to require intensive care for at least 72 hours
* Informed consent obtained from the patient or legal representative

Exclusion Criteria:

* Known pregnancy or breastfeeding
* Participation in another interventional clinical trial within 30 days
* Known immunodeficiency or ongoing immunosuppressive therapy
* Malignancy with life expectancy < 6 months
* Contraindications to focused ultrasound (e.g., splenic trauma, splenectomy, local skin infection)
* Do-not-resuscitate (DNR) order or expected death within 24 hours
* Any other condition deemed unsuitable for participation by the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2025-07-03 (Estimated); Primary Completion 2026-07-02 (Estimated); Study Completion 2026-07-02 (Estimated)

PRIMARY OUTCOMES:
Change in Inflammatory Cytokine Levels | Baseline, Day 3, and Day 5
  Change in plasma levels of key inflammatory cytokines (e.g., TNF-α, IL-1β, IL-6, IL-10) from baseline to Day 3 and Day 5 after randomization.

SECONDARY OUTCOMES:
Change in Lymphocyte Subpopulations | Baseline, Day 3, and Day 5
  Change in plasma levels of key inflammatory cytokines [e.g., CD3⁺T cells (%)、CD3⁺T cells (cells/μL)、CD3-CD19⁺B cells (%)、CD3-CD19⁺B cells (cells/μL)、CD3⁺CD4⁺T cells (%)、CD3⁺CD4⁺T cells (cells/μL)、CD3⁺CD8⁺T cells (%)、CD3⁺CD8⁺T cells (cells/μL)、CD3-(CD16⁺CD56⁺)NK cells (%)、CD3-(CD16⁺CD56⁺)NK cells (cells/μL)] from baseline to Day 3 and Day 5 after randomization.
Change in Organ Function (SOFA Score) | Baseline and Day 5
  Difference in Sequential Organ Failure Assessment (SOFA) scores from baseline to Day 5. The SOFA score ranges from 0 to 24, with higher scores indicating worse organ function and a poorer prognosis.
ICU Length of Stay (LOS) | Through study completion (anticipated average 14 days)
  Duration of ICU hospitalization in days.
28-day mortality rate | 28 days
  All-cause mortality within 28 days after randomization.

IPD SHARING:
Plan to Share IPD: No